CLINICAL TRIAL: NCT06879145
Title: A Randomized, Open, Multicenter Phase II/III Clinical Study of SHR-A2102 for Injection Combined With Adebrelimab (SHR-1316) in Perioperative Treatment of Muscular Invasive Bladder Cancer (MIBC)
Brief Title: Clinical Study on the Treatment of MIBC Patients With SHR-A2102 Injection Combined With Adebrelimab (SHR-1316)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-303
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-02

CONDITIONS: Muscular Invasive Bladder Cancer (MIBC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with SHR-A2102 in combination with a fixed dose of Adebrelimab (Experimental)
  Interventions: Drug: SHR-A2102；Adebrelimab

INTERVENTIONS:
Drug: SHR-A2102；Adebrelimab — Treatment with SHR-A2102 in combination with fixed dose Adebrelimab

SUMMARY:
In phase II, the main objective is to evaluate the efficacy of SHR-A2102 combined with Adebrelimab in the treatment of muscular invasive bladder cancer (MIBC); The main objective of phase III is to evaluate the efficacy of SHR-A2102 for injection combined with Adebrelimab compared with gemcitabine combined with cisplatin in the treatment of muscular invasive bladder cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, gender not limited.
2. The patient voluntarily joined this study and signed informed consent
3. ECOG score is 0 or 1
4. Expected survival period ≥ 2 years.
5. Pathology and imaging diagnosis of non metastatic muscle invasive bladder cancer
6. There are assessable lesions that meet the RECIST 1.1 criteria
7. Enough organ function

Exclusion Criteria:

1. Received systemic anti-tumor therapy 4 weeks before starting the study treatment
2. The toxicity and/or complications of previous anti-tumor treatments have not recovered to NCI-CTCAE ≤ 1 level
3. Subjects known or suspected to have interstitial pneumonia
4. Individuals with any active, known or suspected autoimmune diseases
5. There are clinical symptoms or diseases of the heart that have not been well controlled
6. Diagnosed with any other malignant tumor
7. Subjects who have experienced severe infections within 28 days prior to their first medication use
8. History of immunodeficiency
9. Use of attenuated live vaccine within 28 days prior to the first study medication
10. Have undergone major surgery within 28 days prior to the first administration of medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Phase II: pCR evaluated by researchers; | Three months after the last subject underwent RC+PLD surgery
Phase III: EFS assessed by BICR； | 5 years after the first medication of the last subject

SECONDARY OUTCOMES:
ORR | from first dose to disease progression or death, whichever comes first, up to 3 years
DCR | from first dose to disease progression or death, whichever comes first, up to 3 years
pCR | Three months after MIBC surgery
EFS | from first dose to disease progression or death, whichever comes first, up to 3 years
DFS | from first dose to disease progression or death, whichever comes first, up to 3 years
OS | from first dose to disease progression or death, whichever comes first, up to 3 years
R0 resection rate | One month after the last subject underwent RC+PLD surgery
AE | from Day1 to 90 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided